CLINICAL TRIAL: NCT04640688
Title: Endoscopic Sleeve Gastroplasty / Endoscopic Sleeve Gastroplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 047.GID.2018.D
Record Dates: First submitted 2019-08-12; First posted 2020-11-23 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Bariatric procedures — 510(k) summary K081853 dated June 26, 2008, Endoscopic Sleeve Gastroplasty lecture, Methodist Dallas Medical Center Endobariatric Pathway & Endoscopic Sleeve Gastroplasty Procedure Description

SUMMARY:
This will be a prospective, registry study of an investigational procedure for at least 12 standard of care visits up to 1 year after subject consents for study. Subjects will be enrolled between 8/1/2018 and 8/1/2023. Subjects will undergo a clinically indicated endoscopic procedure and subsequent follow up clinic visits as part of their standard medical care.

Disclaimer: To undergo the procedure there is an out of pocket expense for $9000.

DETAILED DESCRIPTION:
All procedures, barring research activities such as consenting and data collection from Electronic Health Record , will be either clinically indicated and/or standard of care. Subject data will be collected and recorded in a registry which will allow for the prospective review and collection of clinical data related to Endoscopic Sleeve Gastroplasty for safety and efficacy assessment.

Study duration: At least 12 standard of care visits up to 1 year for each subject.

Standard of care follow up visits for Endoscopic Sleeve Gastroplasty are usually 2 weeks, 3 months, 6 months and 12 months post procedure with the physician and 8 follow-up visits over the year with a dietitian. No additional research related visits will be requested. All data will be collected from Electronic Health Record.

Disclaimer: To undergo the procedure there is an out of pocket expense for $9000.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Able to comprehend and provided written informed consent
* Willing to comply with the substantial lifelong dietary restrictions required by the procedure
* History of failure with non-surgical weight-loss methods
* Willing to follow protocol requirements, including providing informed consent, routine follow-up schedule, completing laboratory tests, and completing diet counseling
* Women of childbearing potential ( not post-menopausal or surgically sterilized) must agree to use adequate birth control methods

Exclusion Criteria:

* Below 18 years of age
* Prohibitive anesthetic risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who undergo bariatric procedures at Methodist Dallas Medical Center
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-08-27 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 8/1/2018 and 8/1/2023
  Percentage of total and excess weight loss at 30 days, 3 months, 6 months and 12 months after procedure.

SECONDARY OUTCOMES:
Documentation of safety | 8/1/2018 and 8/1/2023
  procedure readmission rate (in days)

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Kedia, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No